CLINICAL TRIAL: NCT05869305
Title: Efficacy and Safety of Protein Product in Volunteers With Sarcopenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Pornanong Aramwit, Pharm.D., Ph.D, Professor, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: IRBRTA 426/2566
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Soybean Proteins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- whey protein isolate group (Experimental): Whey protein isolate is contained in the sachet.
  Interventions: Dietary Supplement: whey protein isolate
- isolated soy protein group (Experimental): Isolated soy protein, pea protein isolate, and brown rice protein are contained in the sachet.
  Interventions: Dietary Supplement: isolated soy protein
- placebo group (Experimental): Base powder without proteins is contained in the sachet
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: whey protein isolate — Take 1 sachet/day for 12 weeks.
  Arms: whey protein isolate group
Dietary Supplement: isolated soy protein — Take 1 sachet/day for 12 weeks.
  Arms: isolated soy protein group
Dietary Supplement: placebo — Take 1 sachet/day for 12 weeks.
  Arms: placebo group

SUMMARY:
The objective of this study are to evaluate efficacy and safety of protein product in volunteers with sarcopenia.

DETAILED DESCRIPTION:
There are 45 patients in this study. They are randomly divided into 3 groups which are whey protein isolate group, isolated soy protein group, placebo group. They will take the sample 1 sachet/day for 12 weeks. Muscle strength, muscle mass, physical performance, sarcopenia score, body weight, body mass index, protein, immunoglobulins, quality of life, liver function, kidney function, other laboratory value, and adverse effects are evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 20 years
* Sarcopenia score more than 4
* Handgrip strength less than 28 kg in male and less than 18 kg in female and muscle mass less than 7 kg/m2 in male and less than 5.7 kg/m2 in female or Gait speed (6-meter walk) less than 1 m/s
* Can take protein from animal
* Can read and write or have people to look after
* Willing to participate in this study

Exclusion Criteria:

* Allergic to protein from animals and plants
* Hepatitis or cirrhosis
* Glomerular disease or glomerular filtration rate less than 60 ml/min/1.73m2
* Cancer or heart disease
* Cannot walk
* Pregnancy and lactation
* Duodenal surgery
* Take protein supplement within 2 weeks
* Take protein in normal food more than 1.2 g/body weight/day
* Participating in other studies

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-03-20 (Estimated)

PRIMARY OUTCOMES:
Muscle strength | 12 weeks
  Using handgrip strength instrument (high value means high strength)
Muscle mass | 12 weeks
  Using Bioelectrical Impedance Analysis instrument (high value means high mass)
Physical performance | 12 weeks
  Using Gait speed (6-meter walk) (low time period and low score of tired mean high physical performance.
Sarcopenia score | 12 weeks
  Sarcopenia questionnaires (score 1 to 10 means low severity to high severity)
Body weight | 12 weeks
  Body weight of the patients
Body mass index | 12 weeks
  Body mass index of the patients

SECONDARY OUTCOMES:
Nutritional status | 12 weeks
  Nutritional score (score 0 to 17 means lack of nutrition, score 17 to 23.5 means risk to have lack of nutrition, score 24 to 30 means normal nutrition)
Hungry feeling | 12 weeks
  Using visual analogue scale 0 to 10 (No hungry to very hungry)
Quality of life of the patient | 12 weeks
  36-Item Short Form Survey questionnaires shows in quality of life score 0 to 100 (High score means a better outcome)
Concentration of total protein in serum | 12 weeks
  Measure concentration of total protein in serum
Concentration of immunoglobulin in serum | 12 weeks
  Measure concentration of immunoglobulin in serum
Concentration of glucose in serum | 12 weeks
  Measure concentration of glucose in serum
Concentration of calcium in serum | 12 weeks
  Measure concentration of calcium in serum
Concentration of magnesium in serum | 12 weeks
  Measure concentration of magnesium in serum
Concentration of sodium in serum | 12 weeks
  Measure concentration of sodium in serum
Concentration of creatinine in serum | 12 weeks
  Measure concentration of creatinine in serum
Concentration of blood urea nitrogen in serum | 12 weeks
  Measure concentration of blood urea nitrogen in serum
Concentration of aspartate transaminase in serum | 12 weeks
  Measure concentration of aspartate transaminase in serum
Concentration of alanine aminotransferase in serum | 12 weeks
  Measure concentration of alanine aminotransferase in serum
Concentration of alkaline phosphatase in serum | 12 weeks
  Measure concentration of alkaline phosphatase in serum
Skin reaction | 12 weeks
  Found or not found
Respiratory reaction | 12 weeks
  Found or not found
Gastrointestinal tract reaction | 12 weeks
  Found or not found